CLINICAL TRIAL: NCT07042009
Title: inVestigating the effectIveness of nuTritionAl Information Resources for MIlk doNors
Brief Title: Effectiveness of Nutritional Resources for Milk Donors
Acronym: VITAMIN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roehampton (Other)
Collaborators: Countess of Chester NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Dr Simon Dyall, Associate Professor, University of Roehampton
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SD002
Record Dates: First submitted 2025-04-01; First posted 2025-06-27 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Docosahexaenoic Acid Content of the Participants; Docosahexaenoic Acid Content of the Breast Milk
Keywords: omega-3 fatty acids; donor human milk; human milk bank; preterm infants; DHA; docosahexaenoic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nutritional resources (Experimental): Participants in this arm will be provided with the nutritional resources.
  Interventions: Other: Nutritional resources
- Nutritional resources and breast milk DHA content (Experimental): Participants in this arm will be provided with the nutritional resources and feedback on their milk docosahexaenoic acid (DHA) levels
  Interventions: Other: Nutritional resources; Other: Milk docosahexaenoic acid levels
- Control (No Intervention): Participants in this arm will receive standard care.

INTERVENTIONS:
Other: Nutritional resources — The participants will be provided with the nutritional resources only.
  Arms: Nutritional resources; Nutritional resources and breast milk DHA content
Other: Milk docosahexaenoic acid levels — The participants will be provided with information on the levels of docosahexaenoic acid in their breast milk.
  Arms: Nutritional resources and breast milk DHA content

SUMMARY:
Maternal diet influences breast milk nutritional profile; however, a national survey undertaken by the researchers revealed that non-for-profit donor milk banks in the U.K. do not provide specific dietary information to donors. Moreover, the researchers have shown that donor milk in the U.K. provides very low levels of the omega-3 and omega-6 polyunsaturated fatty acids (PUFAs), docosahexaenoic acid (DHA) and arachidonic acid, respectively. These are essential for brain development and immune system function, and preterm infants receiving donor milk do not receive sufficient levels of these nutrients. There is therefore an urgent need to develop nutritional guidelines and resources for milk donors.

Following a systematic review the researchers developed evidence-based nutritional information resources for donors, which would also be applicable more generally to lactating mothers. Those resources were developed in consultation with donors, and healthcare professionals, including dietitians and lactation consultants.

Researchers will evaluate the effectiveness of these resources in terms of acceptance and compliance, and also changes in milk DHA content. The researchers will also assess whether providing feedback on individual's milk DHA content increases milk DHA levels. If successful these resources will be introduced into milk banks across the U.K., and promoted to the wider breastfeeding community.

DETAILED DESCRIPTION:
This is an open label intervention study which lasts eight weeks, but the researchers will operate a rolling recruitment approach, and aim to recruit on average eight participants per month over eight months, to meet the target of 60 participants. Donors will be recruited from the Countess of Chester Hospital milk bank, which is the largest milk bank in England, and typically recruits around 30 to 35 new donors per month, and the researchers are aiming for an approximate 25% conversion rate. At recruitment participants will complete a validated omega-3 polyunsaturated fatty acid (PUFA) Food Frequency Questionnaire (FFQ), provide a bloodspot sample for PUFA analysis, and 1 mL of manually expressed breast milk, which will be expressed at home and brought in by the donors. The bloodspot PUFA analysis will quantify blood docosahexaenoic acid (DHA and eicosapentaenoic acid (EPA) content, which will be used to assess baseline and endpoint participant omega-3 PUFA levels. Then follows the nutritional consultation where the nutritional information resources are provided to the participants. Participants are instructed on how to complete a three-day photo diet diary, to be submitted via a mobile phone application, such as FoodView at the start, middle and end of the study, and how to collect milk drop samples on filter paper. These milk drop samples are collected in weeks 1 and 5, as a drop on a filter paper and posted for analysis. Participants are then randomised so that half will be sent the results of this milk spot analysis, and half will not. After eight weeks there is an endpoint visit, with exit questionnaire and sample collections as at baseline.

The baseline and endpoint milk samples will be manually expressed, and where possible, expressions from more than one time-point on the day will be pooled to allow for differences in milk expression over 24 hours. Samples will be frozen at -70⁰C on the day of expression and shipped on dry ice for analysis. The blood pin prick and drop of breast milk samples will be collected as single drops onto filter paper impregnated with an antioxidant to preserve PUFAs. The paper will be air-dried, wrapped in foil, sealed in polythene bag and stored until analysis. Fatty acids from all samples will be measured by gas chromatography with flame ionisation detector. There is a good correlation between the results of liquid and dried milk spot analysis; however, the dried spot samples are only reported as percentage of total fatty acids and so will primarily be used to provide feedback to the participants. Whereas the liquid milk samples will be reported in absolute amounts as well as percent of the total fatty acids, which allows for a more complete understanding of the composition. Any surplus milk samples will be stored at -70⁰C, where they may be used in future analyses of lipid or nutrient content.

The omega-3 PUFA FFQ will be completed and analysed as per the researchers previous research. For the photo-diet diary, at the initial encounter, each participant will be instructed on how to take the images of foods and beverages over one day. All will use the participants own mobile phone with built-in camera and will use a mobile phone application, such as FoodView. Different meal components will be kept separate on the plate and participants instructed to take one picture per meal. Extra food portions or leftovers are documented by additional pictures. The photo-diaries are taken for two mid-week and one weekend days and submitted via the app for subsequent nutrient analysis using Dietplan software by the research team.

ELIGIBILITY:
Inclusion Criteria:

* New donors from the Countess of Chester Hospital milk bank
* Between six to eight weeks of giving birth

Exclusion Criteria:

* Insufficient comprehension of English to understand the information sheet and consent form and complete the questionnaires
* Currently taking omega-3 PUFA dietary supplements providing greater than 200 mg DHA per day
* Body Mass Index (BMI) ≥30 kg/m2

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Content of omega-3 fatty acids in the participants diet | 8 weeks
  The omega-3 fatty acid content of the participants diet will be assessed from three-day photo-diet diaries taken at the start and end of the study. The participants will use their own mobile phone with a phone application, such as FoodView to record their meals. The omega-3 fatty acid values for alpha-linolenic acid, eicosapentaenoic acid and docosahexaenoic will then be calculated in mg/day from these images using nutrient analysis software, such as Dietplan, and intake levels will be compared between the baseline and endpoint values.

SECONDARY OUTCOMES:
Concentration of docosahexaenoic acid in the participants breast milk | 8 weeks
  The concentration of docosahexaenoic acid in the participants breast milk will be measured by gas chromatography from samples taken at the start and end of the study.
Concentration of omega-3 fatty acids in the participants blood | 8 weeks
  The omega-3 fatty acid concentration of the participants non-fasted blood will be assessed by measuring the docosahexaenoic and eicosapentaenoic acid levels from pin-prick whole-blood samples taken at the start and end of the study. The samples will be analysed by gas chromatography.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Dyall, PhD, Study Chair — University of Roehampton; Yvonne Jeanes, PhD, Study Director — British Dietetic Association

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nessel I, De Rooy L, Khashu M, Murphy JL, Dyall SC. Long-Chain Polyunsaturated Fatty Acids and Lipid Peroxidation Products in Donor Human Milk in the United Kingdom: Results From the LIMIT 2-Centre Cross-Sectional Study. JPEN J Parenter Enteral Nutr. 2020 Nov;44(8):1501-1509. doi: 10.1002/jpen.1773. Epub 2020 Feb 11. PMID 32048312
- [Background] Falize C, Savage M, Jeanes YM, Dyall SC. Evaluating the relationship between the nutrient intake of lactating women and their breast milk nutritional profile: a systematic review and narrative synthesis. Br J Nutr. 2024 Apr 14;131(7):1196-1224. doi: 10.1017/S0007114523002775. Epub 2023 Dec 6. PMID 38053371
- [Background] De Rooy L, Hamdallah H, Dyall SC. Extremely preterm infants receiving standard care receive very low levels of arachidonic and docosahexaenoic acids. Clin Nutr. 2017 Dec;36(6):1593-1600. doi: 10.1016/j.clnu.2016.09.033. Epub 2016 Oct 8. PMID 27756480